CLINICAL TRIAL: NCT00554775
Title: A Randomised Phase II Double Blind Placebo Controlled Trial of Whole Brain Radiotherapy (WBRT) and Tarceva (OSI-774, Erlotinib) in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) With Multiple Brain Metastases [TACTIC]
Brief Title: WBRT & Erlotinib in Advanced NSCLC and Brain Metastases
Acronym: TACTIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IDMC made a recommendation to stop the trial as the target for continuing to the 2nd phase was not met.
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000573254; CRUK-UCL-BRD-05-177; BRD/05/177; EUDRACT-2006-000113-38; CRUK-TACTIC; EU-20792; ISRCTN31916843
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: tumors metastatic to brain; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- erlotinib hydrochloride (Experimental): WBRT plus Tarceva (OSI-774, erlotinib) PO 100 mg daily during WBRT, increasing to 150mg daily after WBRT for up to 24 months
  Interventions: Drug: erlotinib hydrochloride
- placebo (Placebo Comparator): WBRT plus matched placebo for the same schedule and duration as erlotinib hydrochloride arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: erlotinib hydrochloride — PO 100 mg daily during WBRT, increasing to 150mg daily after WBRT for up to 24 months
  Other Names: tarceva; OSI-774
  Arms: erlotinib hydrochloride
Drug: placebo — WBRT plus matched placebo for the same schedule and duration as erlotinib hydrochloride
  Arms: placebo

SUMMARY:
RATIONALE: Radiation therapy uses high energy x-rays to kill tumor cells. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Erlotinib may also make tumor cells more sensitive to radiation therapy. It is not yet known whether giving whole-brain radiation therapy together with erlotinib is more effective than whole-brain radiation therapy alone in treating patients with non-small cell lung cancer and brain metastases.

PURPOSE: This randomized phase II trial is studying whole-brain radiation therapy and erlotinib to see how well they work compared with whole-brain radiation therapy alone in treating patients with advanced non-small cell lung cancer and brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effect of whole-brain radiotherapy (WBRT) and erlotinib hydrochloride vs WBRT alone on neurological progression-free survival at 2 months in patients with advanced non-small cell lung cancer and multiple brain metastases.

Secondary

* Compare the toxicity of these regimens.
* Compare the response rate in these patients.
* Compare quality of life of these patients.
* Compare change in performance status in these patients.
* Compare steroid dosing in these patients.
* Compare sites of progression (cranial or extracranial) in these patients.

OUTLINE: This is a multicenter study. Patients are stratified by presence of extracranial metastases (yes vs no), RTOG recursive partitioning analysis (RPA) score (I vs II) and treatment center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo whole-brain radiotherapy (WBRT) once daily for 5 days. Patients also receive oral erlotinib hydrochloride once daily for up to 24 months.
* Arm II: Patients undergo WBRT as in arm I. Patients also receive oral placebo once daily for up to 24 months.

Quality of life is assessed at baseline, monthly for 12 months, and then at 18 and 24 months.

After completion of study therapy, patients are followed every 1-2 months.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced non-small cell lung cancer (NSCLC) meeting 1 of the following criteria:

  * Newly diagnosed multiple brain metastases not suitable for first-line chemotherapy
  * Relapsed NSCLC with newly diagnosed multiple brain metastases
  * Relapsed after second-line chemotherapy with newly diagnosed multiple brain metastases NOTE: *Biopsy of brain metastases is not required
* Diagnosis of brain metastases must be confirmed by contrast CT scan or MRI within the past 4 weeks

  * Symptoms attributable to brain metastases
  * Patients who have undergone craniotomy with incomplete resection are eligible
* Clinician certain that whole-brain radiotherapy (WBRT) will be beneficial
* No evidence of solitary brain metastasis on MRI that can be treated with surgical resection, radiosurgery, or stereotactic radiotherapy
* No more than 3 sites (organ systems) of extracranial metastases

  * No liver metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* RTOG recursive partitioning analysis (RPA) class I or II
* Serum bilirubin < 2 times upper limit of normal (ULN)
* AST and ALT < 2 times ULN (< 5 times ULN if liver metastases are present)
* Creatinine < 5 times ULN
* Able to take oral medication
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Caretaker able and willing to participate in the study
* Patient and caretaker have access to a telephone and willing to respond to telephone interview
* No other prior or concurrent malignant disease likely to interfere with study treatment or comparisons
* No evidence of other significant laboratory finding or concurrent uncontrolled medical illness, that in the opinion of the investigator, would interfere with study treatment or results comparison or render the patient at high risk for treatment complications including, but not limited to, any of the following:

  * Severe uncontrolled infection
  * Unstable angina
  * Myocardial infarction within the past month
  * Uncontrolled inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)
  * Acute renal failure

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 28 days since prior chemotherapy (for relapsed patients originally treated with chemotherapy)
* No prior cranial radiotherapy
* No prior anti-cancer EGFR therapy (e.g., erlotinib, gefitinib, or cetuximab)
* No prior treatment for brain metastases (e.g., radiosurgery, radiotherapy, or chemotherapy)

  * Prior radiotherapy to the primary tumor and/or systemic treatment to metastatic sites of disease allowed
* No concurrent cyclooxygenase-2 (COX-2) inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Neurological progression-free survival at 2 months | at 2 months

SECONDARY OUTCOMES:
Toxicity | during and for 28 days following Tarceva/placebo treatment.
Response rate | from date of randomisation to radiological progression
Quality of life | completed monthly for the first 12 months and at 18 and 24 months from randomisation
Change in performance status | from baseline
Steroid dosing | from baseline
Sites of progression (cranial or extracranial) | from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Siow M. Lee, MD, PhD, FRCP, Study Chair — University College London Hospitals
Locations (7):
- United Kingdom (7):
  - Charing Cross Hospital, London, England
  - University College of London Hospitals, London, England
  - Christie Hospital, Manchester, England
  - Salisbury District Hospital, Salisbury, England
  - Southampton General Hospital, Southampton, England
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales
  - South West Wales Cancer Institute, Swansea, Wales